CLINICAL TRIAL: NCT06613204
Title: STELLA-FTD: Examination of a Behavior Change Intervention for FTD Family Care Partners
Acronym: STELLA-FTD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Allison Lindauer, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00026023; R01AG084523 (NIH)
Record Dates: First submitted 2024-09-17; First posted 2024-09-25 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Frontotemporal Dementia; Caregiver Burden; Primary Progressive Aphasia (PPA); Corticobasal Syndrome
Keywords: behavioral intervention; FTD
MeSH Terms: conditions — Frontotemporal Dementia; Caregiver Burden; Aphasia, Primary Progressive; Corticobasal Degeneration

STUDY DESIGN:
Intervention Model Description: STELLA-FTD is a 36-week randomized controlled, repeated measures study.
Who Masked: Participant, Care Provider
Masking Description: Care Partners will be randomized to either the test or control group using an electronic randomization process and will be blinded to their group designation. Interventionists will also be blinded to their group designation (test or control) and the differences between the two programs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): Control group, receives information and support in a group setting (N=160 Care Partners).
  Interventions: Behavioral: STELLA-FTD Control
- Test Group (Experimental): Test group, receives information and support in a group setting, but program is different from control (N=160 Care Partners).
  Interventions: Behavioral: STELLA-FTD Test
- Care Recipients with FTD (No Intervention): Care recipients are consented to inform them of their rights, but they do not take part in any activities (N=320 Care Recipients).

INTERVENTIONS:
Behavioral: STELLA-FTD Control — Participants receive information about FTD and support via weekly group video-conference-based meetings.
  Arms: Control Group
Behavioral: STELLA-FTD Test — The test group receives a information and support, but with a focus that is different from the Control Group
  Arms: Test Group

SUMMARY:
The purpose of this nationwide study is to test STELLA-FTD (Support via Telehealth: Living and Learning with Advancing Alzheimer's Disease)-FTD, an intervention to specifically address the needs of family Care Partners of persons with frontotemporal degeneration (FTD). STELLA-FTD is a multicomponent videoconference-based intervention designed to facilitate effective use of community and peer resources to foster effective management of behavioral and psychological symptoms of dementia. The study is recruiting families from across the United States.

DETAILED DESCRIPTION:
The study will enroll a total sample of up to 640 participants: 320 family Care Partners and their 320 Care Recipients with FTD. For our study "family Care Partner" includes any person who is considered "family" to the person with FTD, such as direct relations, fictive kin, close friends and neighbors. "Care Recipient" is defined as an individual with an FTD diagnosis noted by the AFTD: bv-FTD, PPA, progressive supranuclear palsy (PSP), corticobasal degeneration (CBD), or ALS with FTD. Care Recipients with FTD will not participate in intervention but will be consented (and thus enrolled) because data will be collected about them. The study will test to see if our program helps Care Partners.

The STELLA-FTD intervention is delivered over 8 sessions within 10 consecutive weeks in 1-hour "live" video-based group sessions led by two guides. There will be two intervention groups, the control group and the test group. There will be up to 8 Care Partners per group, which allows for the development of mutual trust and commitment.

Care Partners will be randomized to either the test or control group using an electronic randomization process and will be blinded to their group designation. Both groups will receive information and support (via videoconferencing). The test group will receive a different program than the control group. Care Partners will fill out 6 long surveys while in the study, and a brief weekly survey.

ELIGIBILITY:
Inclusion Criteria: Family Care Partner

* Adult caring for family member with FTD.
* Provides 4 or more hours of care/week. Does not have to reside with.
* Identifies at least 2 moderately upsetting behaviors in the person with FTD.
* Speaks and understands English to be able to participate in intervention.
* Owns a telephone (smartphone, cell phone or landline).
* Has email and mailing address to receive computer, study materials and surveys.
* Provides informed consent to participate in the research.
* Lives in the US

Inclusion Criteria: Person with FTD

* Diagnosis of FTD
* Family member of a Care Partner (this can be a relative, spouse, or close kin that is considered family).
* Lives in US

Exclusion Criteria: Person with FTD

* No Frontotemporal Degeneration diagnosis.
* Unable to leave Care Partner during STELLA-FTD sessions.
* Enrolled in hospice.

Exclusion Criteria: Family Care Partner

* Unable to find activity for Care Recipient during STELLA-FTD sessions to allow Care Partner to work privately with Guide and other Care Partners.
* Hearing and/or vision problems severe enough to prevent participation.
* Refuses to be video-recorded during STELLA-FTD sessions.
* Unwilling or unable to adequately follow study instructions and participate in study procedures.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Revised Memory and Behavior Problems Checklist, Frequency, Original Scale | 1 month pre-intervention; 1 week pre-intervention, 4 weeks after intervention start; 8 week post intervention; 2 and 6 months post intervention
  Efficacy will be assessed by measuring pre/post changes on the RMBPC. The RMBPC is a 24-item caregiver report measure, 5-point Likert scale with higher scores on frequency indicate more upsetting behaviors Frequency range is 0 (never occurred) to 4 (daily or more often). Frequency score range is 0 to 96
Revised Memory and Behavior Problems Checklist, Reactivity, Original Scale | 1 month pre-intervention; 1 week pre-intervention, 4 weeks after intervention start; 8 week post intervention; 2 and 6 months post intervention
  Efficacy will be assessed by measuring pre/post changes on the RMBPC. The RMBPC is a 24-item caregiver report measure, 5-point Likert scale with higher scores on reactivity indicate more Care Partner burden. Frequency range is 0 (no burden) to 4 (high burden). Frequency score range is 0 to 96

SECONDARY OUTCOMES:
Self-efficacy for symptom management and support service use | 1 month pre-intervention; 1 week pre-intervention, 8 week post intervention; 2 and 6 months post intervention
  10-item scale to measure self-efficacy. Assesses caregiver certainty that they will use services and support programing. 1= not at all certain, to 10=very certain. Scores range from 10 to 100, with 100 being high certainty.
Neuropsychiatric Inventory-Caregiver Self-efficacy Scale | 1 month pre-intervention; 1 week pre-intervention, 8 week post intervention; 2 and 6 months post intervention
  Measures frequency of behaviors related to frontotemporal dementia and Care Partner confidence in managing behaviors. Frequency is rated on a scale of 1 (occasionally) to 4 (very frequently), severity is rated from 1 (mild) to 3 (severe), and caregiver distress is rated from 0 (no distress) to 5 (extreme or very severe). Total scores are calculated by multiplication of the frequency and severity for each symptom and the addition of all item scores, with a range of 0-144. The distress score total is calculated by the sum of all the individual domain scores, with a range of between 0 and 60. If a behavioral symptom is noted, the care partner is asked to about how confident they are in addressing it, Responses range from 4 (not at all confident), 3 (fairly confident), 2 (confident), and 1 (very confident).
Preparedness for Caregiving Scale | 1 month pre-intervention; 1 week pre-intervention, 8 week post intervention; 2 and 6 months post intervention
  10-item measure that assesses how prepared care partners feel to care for their family member with dementia. Ranges from 0 (not at all prepared) to 40 (very well prepared).
Personalized Target Behavior Survey | 1 week pre-intervention, 8 week post intervention
  On STELLA-FTD Website, measures frequency and reactivity of up to 3 personalized behaviors identified by Care Partners. Care partners rate how often the 5-point Likert scale with higher scores on frequency indicate more upsetting behaviors Frequency range is 0 (never occurred) to 4 (daily or more often). Frequency score range is 0 to 4 for each Target behavior. Higher scores indicate higher frequency and burden.
Service and Support use survey | 1 month pre-intervention; 1 week pre-intervention, 8 week post intervention; 2 and 6 months post intervention
  10-item survey that queries participants about service use. Score is not on a scale.
Support via Telehealth: Living and Learning with Advancing Frontotemporal Dementia Experience Survey | 1 week post intervention
  18-item- survey on satisfaction, privacy, ease of use. Scores range from 1 (strongly disagree) to 5 (strongly agree). Total score ranged 18-90, higher scores are better
Orbit Survey | Weekly, starts at Week 1, ends after week 36.
  Weekly survey of burden, service use, medication use. Score is not on a scale.
Revised Memory and Behavior Problem Checklist Frontotemporal Degeneration Supplement, Frequency | 1 month pre-intervention; 1 week pre-intervention, 4 weeks after intervention start; 8 week post intervention; 2 and 6 months post intervention
  Measures frequency of upsetting frontotemporal behaviors. 9 items, scores range from 0 (no behaviors) to 36 (all behaviors)
Revised Memory and Behavior Problem Checklist Frontotemporal Degeneration Supplement, Reactivity | 1 month pre-intervention; 1 week pre-intervention, 4 weeks after intervention start; 8 week post intervention; 2 and 6 months post intervention
  Measures caregivers reactions to upsetting frontotemporal behaviors. 9 items, scores range from 0 (no reactivity) to 36 (high reactivity)
Clinical Dementia Rating Scale plus Frontotemporal Lobar Degeneration | One time assessment at enrollment
  This is an 8-item survey that assesses disease severity, with 0=no impairment to 3=severe impairment. Range is 0-24 (Sum of boxes)
Ten Item Personality Inventory | Once, at Week 1 of intervention
  10 items that assess personality type. Respondents note how they agree with each. personality type, from
  1=Disagree strongly 2 = Disagree moderately 3 = Disagree a little 4 = Neither agree nor disagree 5 = Agree a little 6 = Agree moderately 7 = Agree strongly
  Score is not on a scale.
Contact Survey | Week 13, 20, and 36
  Nine questions query caregivers about if they contacted other caregivers in the study, and, if so, how often. Score is not on a scale

CONTACTS AND LOCATIONS:
Overall Officials: Allison Lindauer, PhD, APRN, Principal Investigator — Oregon Health and Science University; Aimee Mooney, MA, CCC-SLP, Study Director — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Aggregated data for journal articles and presentations, IPD via data request to OHSU
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 2/15/2025-7/14/2029
Access Criteria: Scientists can contact our center to request data
URL: https://www.ohsu.edu/alzheimers-disease-research-center/data-resources

REFERENCES:
- [Background] Lindauer A, Smith S, Gothard S, Mattek N, Tran L, Mooney A. 'There's no straight line...' a consumer-informed intervention for FTD family care partners: the STELLA-FTD pilot study. Aging Ment Health. 2023 Sep-Oct;27(10):2000-2010. doi: 10.1080/13607863.2023.2250741. Epub 2023 Sep 1. PMID 37655616
- Available data/document: data set — http://www.ohsu.edu/alzheimers-disease-research-center/data-resources